CLINICAL TRIAL: NCT04982393
Title: BONAPH1DE, A Prospective Observational Study of Patients With Primary Hyperoxaluria Type 1 (PH1)
Acronym: BONAPH1DE
Status: Active, not recruiting | Type: Observational
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: ALN-GO1-007
Record Dates: First submitted 2021-07-20; First posted 2021-07-29 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Primary Hyperoxaluria Type 1
Keywords: PH1; Lumasiran; Primary Hyperoxaluria Type 1
MeSH Terms: conditions — Primary hyperoxaluria type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with PH1: Patients with a diagnosis of PH1 will be eligible for the study and will be managed and treated per routine clinical practice.

SUMMARY:
The purpose of this study is to describe the natural history and progression of patients diagnosed with PH1, and to characterize the long-term real-world safety and effectiveness of lumasiran.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of PH1, per physician's determination

Exclusion Criteria:

* Currently enrolled in a clinical trial for any investigational agent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with PH1 will be managed and treated per routine clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events in Lumasiran Treated Patients | Up to 7 years

SECONDARY OUTCOMES:
Incidence of Selected Events of Interest in PH1 Patients | Up to 7 years
  Selected events of interest are defined as hepatic events, kidney stones, acute kidney injury events, nephrocalcinosis, chromic kidney disease, kidney failure, and any cardiac, bone, skin, eye, hematological, or neuropathic manifestations due to oxalosis.
12-Item Short Form Health Survey Version 2 (SF-12 V2) (Standard Version) | Up to 7 years
  SF-12 V2 is a 12-question measure capturing global quality of life and overall health status and evaluates the following 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional, and mental health.
Change in Urinary Oxalate Excretion | Baseline and every 12 months for up to 7 years
Change in Plasma Oxalate | Baseline and every 12 months for up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Alnylam Pharmaceuticals
Locations (30):
- United States (8):
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Rochester, Minnesota
  - Clinical Trial Site, Cincinnati, Ohio
  - Clinical Trial Site, Pittsburgh, Pennsylvania
  - Clinical Trial Site, Dallas, Texas
  - Clinical Trial Site, Houston, Texas
- Belgium (2):
  - Clinical Trial Site, Ghent
  - Clinical Trial Site, Liège
- Canada (3):
  - Clinical Trial Site, Hamilton, Ontario
  - Clinical Trial Site, Toronto, Ontario
  - Clinical Trial Site, Laurier, Quebec
- France (3):
  - Clinical Trial Site, Bordeaux
  - Clinical Trial Site, Lyon
  - Clinical Trial Site, Paris
- Germany (3):
  - Clinical Trial Site, Berlin
  - Clinical Trial Site, Cologne
  - Clinical Trial Site, Hamburg
- Clinical Trial Site, Jerusalem, Israel
- Italy (3):
  - Clinical Trial Site, Orbassano, Torino
  - Clinical Trial Site, Milan
  - Clinical Trial Site, Verona
- Clinical Trial Site, Amsterdam, Netherlands
- Spain (3):
  - Clinical Trial Site, Santa Cruz de Tenerife, Canary Islands
  - Clinical Trial Site, Barcelona
  - Clinical Trial Site, Las Palmas
- Clinical Trial Site, Bern, Switzerland
- United Kingdom (2):
  - Clinical Trial Site, London, England
  - Clinical Trial Site, London

IPD SHARING:
Plan to Share IPD: No